CLINICAL TRIAL: NCT00389038
Title: Drug and Non-Drug Treatment of Pediatric Chronic Headache
Brief Title: Pediatric Chronic Headache Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Scott W. Powers, PhD ABPP FAHS, Professor, Co-Director of the Headache Center, Cincinnati Children's Hospital Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01NS050536 (NIH); 1R01NS050536-01A1 (NIH)
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Headache
Keywords: headache; coping skills training; amitriptyline; attention control
MeSH Terms: conditions — Headache | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping Skills Training + Amitriptyline (Active Comparator): Behavioral coping skills training--Behavioral Treatment session 1 and 2: Doses are one session a week for 8 weeks, followed by one session a month for 2 months, followed by 1 session every three months for 1 year.
  Interventions: Behavioral: Coping Skills Training; Drug: Amitriptyline
- Headache Education + Amitriptyline (Active Comparator): Behavioral headache education
  Interventions: Behavioral: Headache Education; Drug: Amitriptyline

INTERVENTIONS:
Behavioral: Coping Skills Training — Behavioral Treatment 1 (coping skills training)--Behavioral Treatment session 1 and 2: Doses are one session a week for 8 weeks, followed by one session a month for 2 months, followed by 1 session every three months for 1 year.
  Arms: Coping Skills Training + Amitriptyline
Behavioral: Headache Education — Behavioral Treatment 2 (headache education)
  Arms: Headache Education + Amitriptyline
Drug: Amitriptyline — Amitriptyline: up to 1 mg/kg capsule taken once daily at bedtime. Taken up to Week 20. After Week 20 medications and doses may change with standard care.

SUMMARY:
The purpose of this trial is to evaluate the efficacy of combined behavioral and pharmacological treatment on chronic daily headache in children ages 10 to 17.

DETAILED DESCRIPTION:
Chronic daily headache (CDH)--defined as having headaches 15 or more days per month--is a frequent and debilitating condition in children that results in severe decreased quality of life and emotional stress. Very little is known about the most effective types of treatment for CDH in children and adolescents. Development of effective interventions for youth with CDH could potentially prevent the progression of a very painful and costly condition into adulthood. Treatments combining pharmacological (drug) interventions with behavior change have been found effective in treating adults with chronic pain, including headaches, but have been understudied in children.

The goal of this randomized, controlled clinical trial is to determine the efficacy of combined behavioral and drug treatment of CDH in youth ages 10 to 17. In the study, scientists will investigate if a combination of pain coping skills training (CST) and the drug amitriptyline (AMI)--CST-AMI--is effective in reducing headache frequency, functional disability, and symptoms of depression. More specifically, the researchers will evaluate if CST-AMI is superior to AMI combined with an attention control (ATT). The CST will mainly focus on learning skills for coping with pain, and the ATT will focus on understanding chronic headaches and lifestyle information.

Participants will be randomly assigned to one of the two treatment groups: CST-AMI or ATT-AMI. Those assigned to CST-AMI will complete 8 weekly sessions of coping training and 2 monthly maintenance-promoting sessions. Sessions will focus on teaching biofeedback, muscle relaxation techniques, imagery, distraction, activity pacing, problem solving, and calming techniques, using a treatment manual developed and tested in youth with CDH. Those assigned to ATT-AMI will receive the same amount of therapist support and attention but not the active behavioral training. All participants will receive the study medication, AMI.

Headache frequency, functional disability, pain and headache characteristics, quality of life, and symptoms of depression will be assessed before and after treatment, and reassessed at 3, 6, 9, and 12 months. For participants, duration of the study--which includes treatment and follow-up phases--lasts about 18 months. The treatment phase includes 12 study visits and the follow-up phase includes 4 study visits.

The long-term objective of this research is to establish effective treatments for CDH in youth that lead to significantly reduced headache frequency and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic daily headache based on definition of 15 or more headache days per month measured by a prospective daily headache diary
* females or males between the ages of 10-17
* PedMIDAS Disability Score > 20, indicating at least moderate disruption in daily activities

Exclusion Criteria:

* medication overuse as defined in the ICHD-II criteria (NSAID or other simple analgesic on ≥ 15 days/ month for >3 months; triptan intake in any formulation ≥ 10 days/month on a regular basis of ≥ 3 months)
* current treatment with amitriptyline
* no other current prophylactic antimigraine medication within a period equivalent to < 5 half-lives of that medication before entering the screening phase
* other chronic pain condition such as juvenile primary fibromyalgia syndrome, complex regional pain syndrome-II
* abnormal findings on EKG
* current or past history of severe orthostatic intolerance or severe levels of orthostatic dysregulation (orthostatic hypotension or postural orthostatic tachycardia syndrome)
* significant documented developmental delay or impairments such as autism, cerebral palsy or mental retardation
* present or lifetime psychiatric diagnosis that meets DSM-IV criteria for bipolar disorder, major depressive disorder or psychosis
* PedMIDAS Disability Score of > 140, indicating need for multi-systemic therapies to address very significant level of disability
* youth who are pregnant, or those females who are sexually active and not using a medically accepted form of contraception (barrier or hormonal methods) or do not agree to be abstinent during the study
* disallowed medications/products: opioids, antipsychotics, antimanics, barbiturates, benzodiazepines, muscle relaxants, sedatives, tramadol

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2006-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Headache diaries assess headache frequency. | Completed one month prior to first visit, then weekly up to Week 20, then one month prior to Month 3, 6, 9, and 12 Follow-Up Visits.

SECONDARY OUTCOMES:
The Child Depression Inventory. | Completed at Baseline, Week 20, and Months 3, 6, 9, and 12.
The PedsQL measures the impact of chronic illness and quality of life. | Completed at Baseline, Week 20, and Months 3, 6, 9, and 12.
Pediatric Migraine Disability Assessment (PedMIDAS) evaluates the impact of headaches on life activities. | Completed at Baseline, Week 20, and Months 3, 6, 9, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Scott W. Powers, PhD, ABPP, FAHS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, 3333 Burnet Avenue, Mail Location 3015, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Rettig EK, Ergun G, Warfield JR, Slater SK, LeCates SL, Kabbouche MA, Kacperski J, Hershey AD, Powers SW. Predictors of Improvement in Pediatric Chronic Migraine: Results from the Cognitive-Behavioral Therapy and Amitriptyline Trial. J Clin Psychol Med Settings. 2022 Mar;29(1):113-119. doi: 10.1007/s10880-021-09782-4. Epub 2021 May 24. PMID 34028656
- [Derived] Kroner JW, Peugh J, Kashikar-Zuck SM, LeCates SL, Allen JR, Slater SK, Zafar M, Kabbouche MA, O'Brien HL, Shenk CE, Kroon Van Diest AM, Hershey AD, Powers SW. Trajectory of Improvement in Children and Adolescents With Chronic Migraine: Results From the Cognitive-Behavioral Therapy and Amitriptyline Trial. J Pain. 2017 Jun;18(6):637-644. doi: 10.1016/j.jpain.2017.01.002. Epub 2017 Jan 18. PMID 28108386
- [Derived] Kroner JW, Hershey AD, Kashikar-Zuck SM, LeCates SL, Allen JR, Slater SK, Zafar M, Kabbouche MA, O'Brien HL, Shenk CE, Rausch JR, Kroon Van Diest AM, Powers SW. Cognitive Behavioral Therapy plus Amitriptyline for Children and Adolescents with Chronic Migraine Reduces Headache Days to </=4 Per Month. Headache. 2016 Apr;56(4):711-6. doi: 10.1111/head.12795. Epub 2016 Mar 18. PMID 26992129
- [Derived] Powers SW, Kashikar-Zuck SM, Allen JR, LeCates SL, Slater SK, Zafar M, Kabbouche MA, O'Brien HL, Shenk CE, Rausch JR, Hershey AD. Cognitive behavioral therapy plus amitriptyline for chronic migraine in children and adolescents: a randomized clinical trial. JAMA. 2013 Dec 25;310(24):2622-30. doi: 10.1001/jama.2013.282533. PMID 24368463
- [Derived] Zafar M, Kashikar-Zuck SM, Slater SK, Allen JR, Barnett KA, Lecates SL, Kabbouche MA, Hershey AD, Powers SW. Childhood abuse in pediatric patients with chronic daily headache. Clin Pediatr (Phila). 2012 Jun;51(6):590-3. doi: 10.1177/0009922811407181. Epub 2011 May 18. No abstract available. PMID 21593054
- See also: Cincinnati Children's Hospital Lab Web Page — http://www.cincinnatichildrens.org/research/div/psychology/faculty-labs/powers/